CLINICAL TRIAL: NCT06040320
Title: A Phase I/II Study of Frontline Therapy With Polatuzumab Vedotin (Pola) Plus Rituximab (R) in Patients With Post-transplant Lymphoproliferative Disorder (PTLD)
Brief Title: Polatuzumab Vedotin (Pola) Plus Rituximab (R) in Patients With Post-transplant Lymphoproliferative Disorder (PTLD)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202308116
Record Dates: First submitted 2023-09-09; First posted 2023-09-15 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Post-transplant Lymphoproliferative Disorder
Keywords: PTLD; Non-Hodgkin's lymphoma; Risk stratification; Front-line
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — polatuzumab vedotin; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Polatuzumab vedotin + Rituximab (Safety Lead-in Low Risk/Interim Complete Remission) (Experimental): * Cycle 1 (21 days)
    * Day 1: polatuzumab vedotin + rituximab
    * Day 8: rituximab
    * Day 15: rituximab
  * Cycle 2 (21 days)
    * Day 1: polatuzumab vedotin + rituximab
  * After Cycle 2, a response assessment will be performed. Patients who show a complete response (and are therefore determined to be low risk) will continue to receive polatuzumab vedotin + rituximab on Day 1 of each 21-day cycle for 4 additional cycles (6 cycles of treatment total).
  Interventions: Drug: Polatuzumab vedotin; Drug: Rituximab
- Polatuzumab vedotin + Rituximab (Expansion Low Risk/Interim Complete Remission) (Experimental): * Cycle 1 (21 days)
    * Day 1: polatuzumab vedotin + rituximab
    * Day 8: rituximab
    * Day 15: rituximab
  * Cycle 2 (21 days)
    * Day 1: polatuzumab vedotin + rituximab
  * After Cycle 2, a response assessment will be performed. Patients who show a complete response (and are therefore determined to be low risk) will continue to receive polatuzumab vedotin + rituximab on Day 1 of each 21-day cycle for 4 additional cycles (6 cycles of treatment total).
  Interventions: Drug: Polatuzumab vedotin; Drug: Rituximab
- Polatuzumab vedotin + Rituximab + CHP (Safety Lead-in High Risk/Lack of Interim Complete Remission)) (Experimental): * Cycle 1 (21 days)
    * Day 1: polatuzumab vedotin + rituximab
    * Day 8: rituximab
    * Day 15: rituximab
  * Cycle 2 (21 days)
    * Day 1: polatuzumab vedotin + rituximab
  * After Cycle 2, a response assessment will be performed. Patients who show anything other than a complete response (and are therefore determined to be high risk) will receive polatuzumab vedotin + rituximab + CHP (cyclophosphamide + doxorubicin + prednisone) on Day 1 of each 21-day cycle for 4 additional cycles, followed by 2 final cycles of CHP alone on Day 1 (8 cycles of treatment total).
  Interventions: Drug: Polatuzumab vedotin; Drug: Rituximab; Drug: CHP
- Polatuzumab vedotin + Rituximab + CHP (Expansion High Risk/Lack of Interim Complete Remission) (Experimental): * Cycle 1 (21 days)
    * Day 1: polatuzumab vedotin + rituximab
    * Day 8: rituximab
    * Day 15: rituximab
  * Cycle 2 (21 days)
    * Day 1: polatuzumab vedotin + rituximab
  * After Cycle 2, a response assessment will be performed. Patients who show anything other than a complete response (and are therefore determined to be high risk) will receive polatuzumab vedotin + rituximab + CHP (cyclophosphamide + doxorubicin + prednisone) on Day 1 of each 21-day cycle for 4 additional cycles, followed by 2 final cycles of CHP alone on Day 1 (8 cycles of treatment total).
  Interventions: Drug: Polatuzumab vedotin; Drug: Rituximab; Drug: CHP

INTERVENTIONS:
Drug: Polatuzumab vedotin — Given at 1.8 mg/kg
  Other Names: Polivy
Drug: Rituximab — Given at 375 mg/m^2
  Other Names: Rituxan
Drug: CHP — Cyclophosphamide (750 mg/m^2) + doxorubicin (50 mg/m^2) + prednisone (100 mg days 2-6)
  Arms: Polatuzumab vedotin + Rituximab + CHP (Expansion High Risk/Lack of Interim Complete Remission); Polatuzumab vedotin + Rituximab + CHP (Safety Lead-in High Risk/Lack of Interim Complete Remission))

SUMMARY:
This study will test polatuzumab vedotin in combination with rituximab in patients with treatment-naïve CD20-positive post-transplant lymphoproliferative disorder (PTLD) based on the established efficacy of polatuzumab vedotin in B-cell lymphomas and the inadequate response rate of PTLD to single-agent rituximab. The hypothesis is that this combination therapy will be safe, well-tolerated, and effective. If so, patients with PTLD will be able to be spared the toxicity of anthracycline-based chemotherapy. Additionally, the role of the tumor microenvironment and the role of anellovirus, a non-human pathogen virus, will be explored as prognostic markers in PTLD.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated biopsy-confirmed CD20-positive monomorphic post-transplant lymphoproliferative disorder (or CD20-positive lymphoma associated with immune deficiency) arising after solid organ or hematopoietic stem cell transplant. This may be defined by either the 2016 World Health Organization classification of lymphoid neoplasms or the 2022 International consensus Classification of Mature Lymphoid Neoplasms or the 2022 World Health Organization classification.
* At least 18 years of age.
* ECOG performance status ≤ 3.
* Adequate hematologic and organ function (unless due to underlying lymphoma per the investigator) as defined below:

  * Absolute neutrophil count ≥ 1.0 K/cumm
  * Platelets ≥ 75 K/cumm
  * Hemoglobin ≥ 8.0 g/dL
  * Total bilirubin < 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) < 2.5 x IULN
  * Creatinine clearance > 30 mL/min measured or by Cockcroft-Gault
* Note: Patients with extensive bone marrow involvement by lymphoma and/or disease-related cytopenias may be enrolled if the following criteria are met:

  * ANC ≥ 0.5 K/cumm
  * Platelets ≥ 50 K/cumm
  * Hemoglobin ≥ 7.0 g/dL
* The effects of polatuzumab vedotin and rituximab on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a participant become pregnant or suspect pregnancy while participating in this study, the participant must inform the treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document.

Exclusion Criteria:

* Active central nervous system involvement with lymphoma / PTLD.
* Current grade ≥ 2 peripheral neuropathy.
* Current ejection fraction < 40% on transthoracic echocardiogram or multigated acquisition (MUGA) scan
* Subjects with history of concurrent second cancers requiring active, ongoing systemic treatment with the following exceptions:

  * Patients with non-melanoma skin cancer or carcinoma in situ of the cervix will not be excluded.
  * Patients with previous malignancies are eligible if disease-free for > 2 years.
  * Patients on long term hormonal therapy to prevent recurrence of a prior cancer (e.g., hormonal therapy for breast cancer) will not be excluded.
* Currently receiving any other investigational agents or received any investigational agents during the 4 weeks prior to the first dose of polatuzumab vedotin.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to polatuzumab vedotin, rituximab, or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (bacterial, fungal, viral, parasitic, or mycobacterial), interstitial lung disease, active non-infectious pneumonitis, congestive heart failure NYHA grade ≥ 3, unstable angina pectoris, or cardiac arrhythmia.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to C1D1
* Patients with HIV are eligible provided the meet the following criteria:

  * On antiretroviral regimen and stable on that regimen
  * Healthy from an HIV perspective
  * CD4 count > 250 cells/mcL
  * Minimal anticipated interactions or overlapping toxicity with polatuzumab vedotin or rituximab
  * HIV viral load < 200 copies/mm3 by standard clinical assays
* Active hepatitis B infection.

  * Patients who are hepatitis B surface antigen (HBsAg) negative and hepatitis B core antibody (HBcAb) positive must be negative for hepatitis B virus (HBV) polymerase chain reaction (PCR) to be eligible for study participation.
* Active hepatitis C infection.

  * Patients who are positive for hepatitis C virus (HCV) antibody must be negative for HCV by PCR to be eligible for study participation.
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study, or which could affect compliance with the protocol or interpretation of results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-10-04 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2032-05-31 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of treatment-related adverse events (AEs) | From start of treatment through 30 days after completion of treatment (estimated to be 5-7 months)
Number of dose-limiting toxicities (DLTs) (Safety Lead-In Cohort only) | From start of treatment through cycle 2 (estimated to be 42 days, each cycle is 21 days)
  A dose-limiting toxicity (DLT) is defined as an occurrence of an adverse event delineated by the protocol that is at least possibly related to polatuzumab vedotin, rituximab, or the combination within Cycle 1 or Cycle 2.
Rate of completion of the regimen | Through completion of treatment (estimated to be 4-6 months)

SECONDARY OUTCOMES:
Complete metabolic response (CR) rate by PET/CT | After cycle 2 (estimated to be day 42, each cycle is 21 days)
  -Per Lugano Response Criteria
Complete metabolic response (CR) rate by PET/CT | End of treatment (estimated to be between 4-6 months)
  -Per Lugano Response Criteria
Overall response rate (ORR) | End of treatment (estimated to be between 4-6 months)
  * Per Lugano Response Criteria
  * Overall Response Rate: The proportion of patients who have a complete or partial response to therapy.
Best overall response | Through completion of treatment (estimated to be between 4-6 months)
  * Per Lugano Response Criteria
  * Best Overall Response: Best response recorded from start of treatment until disease progression/recurrence (taking as reference for PD the smallest measurements recorded since the treatment started).
Duration of response | Through 5 years from completion of treatment (estimated to be between 64 and 66 months)
  * Per Lugano Response Criteria
  * Duration of Response: The time from onset of response to disease progression or death in patients who achieve complete or partial response.
Progression-free survival (PFS) | Through 5 years from completion of treatment (estimated to be between 64 and 66 months)
  * Per Lugano Response Criteria
  * Progression-Free Survival: The time from initiation of treatment to the occurrence of disease progression or death.
Overall survival (OS) | Through 5 years from completion of treatment (estimated to be between 64 and 66 months)
  -Overall Survival: The time from initiation of treatment to death.

CONTACTS AND LOCATIONS:
Overall Officials: Neha Mehta-Shah, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu